CLINICAL TRIAL: NCT02195518
Title: A Multi-centre, Single-arm, Open-label Study to Evaluate the Efficacy and Safety of Tenofovir Disoproxil Fumarate(TDF) Treatment in Chinese Chronic Hepatitis B (CHB) Subjects Following Failure of Multiple Nucleos(t)Ide Analogues(NAs)
Brief Title: Tenofovir Disoproxil Fumarate (TDF) 300mg 3 Years RD Therapy Chinese Chronic Hepatitis B (CHN) CHB Multiple Nucleos(t)Ide Analogues (NAs) Failure Points Pts PH4 PMS Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201215
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic Hepatitis B; Tenofovir disoproxil fumarate; Failure of multiple NAs treatment
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tenofovir Disoproxil Fumarate (Experimental): All enrolled subjects will receive open label TDF at a dose of 300 milligram (mg) orally once daily during the study period.
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — Tenofovir disoproxil fumarate tablets supplied will be white, almond-shaped, film-coated tablets containing 300 mg of TDF. Each tablet contains the following inactive ingredients: microcrystalline cellulose, lactose monohydrate, pregelatinised starch, croscarmellose sodium, and magnesium stearate.

SUMMARY:
This is a phase IV, single-arm, open-label, multi-centre study to assess the efficacy of TDF in Chronic hepatitis B (CHB) subjects following failure of multiple Nucleos(t)ide analogues (NAs). The study will enrol 200 CHB subjects following failure of multiple NAs. Subjects will be assessed for eligibility at a screening visit, with eligible subjects returning for a baseline assessment after approximately 4 weeks (Screening phase). In the treatment phase all enrolled subjects will receive open label TDF at a dose of 300 milligrams (mg) orally once daily. All the eligible study subjects will undergo safety and efficacy assessments every 12 weeks for a total of 14 visits. Tenofovir disoproxil fumarate, the oral pro-drug of tenofovir (TFV), is a nucleotide analogue that inhibits viral polymerases by direct binding and after incorporation into deoxyribonucleic acid (DNA), by termination of the DNA) chain. TDF is a highly potent treatment in treatment-naïve and lamivudine (LAM) resistant CHB patients. The purpose of our study is to evaluate the efficacy of TDF treatment in Chinese CHB patients following failure of multiple NAs. In addition, the study will also explore the relationship of baseline factors and early HBV DNA suppression to long-term virological response. The efficacy of TDF in multi-drug resistant patients will be analysed separately. The data generated by this study could then be used to optimize the clinical application of TDF and provide new evidence for management of the HBV infections following failure of multiple NAs. The result of this study will help Chinese physicians better manage the CHB patients following failure of multiple NAs.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65years (inclusive). Male or female; a female is eligible to enter and participate in this study if she is of: Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
* Child-bearing potential, has a negative serum pregnancy test at baseline, and agrees to one of the following methods for avoidance of pregnancy during the period of the study and until 30 days after last dose of study medication: Oral contraceptive, either combined or progestogen alone, Injectable progestogen, Implants of levonorgestrel, Oestrogenic vaginal ring, Percutaneous contraceptive patches., Intrauterine device (IUD) or intrauterine system (IUS) showing that the expected failure rate is less than 1% per year as stated in the IUD or IUS product label, Has a male partner who is sterilised, Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film /cream/suppository).
* The ability to understand and sign a written informed consent prior to any study-related procedure and comply with the requirements of the study.
* Positive HBsAg for more than 6 months, and anti-HBs negative.
* Serum HBV DNA level >=200 IU/mL at study screening (Use central lab results).
* Experienced multiple NAs treatment failure which is defined as HBV DNA greater than 200 IU/mL after at least two NAs treatment (at least 6 months continuous treatment for each NA(s), total duration is no less than 12 months). In addition, subjects judged by the treating physician to have adhered to previous NA therapy.
* Agreement not to participate in any other investigational trials or to undertake other HBV systemic antiviral or interferon (IFN) regimens during participation in this study.

Exclusion Criteria:

* Hepatocellular carcinoma as evidenced by one of the following: Suspicious foci on ultrasound or radiological examination, Normal ultrasound but a history of rising serum alpha-fetoprotein and serum alpha-fetoprotein >20 nanogram (ng) per mL at screening.
* Clinical signs of decompensated liver disease at baseline. These may include but are not limited to:Total serum bilirubin >1.5 x Upper limit of the normal range (ULN), International Normalized Ratio >1.3, Serum albumin <32grams per Liter (g/L), History of clinical hepatic decompensation (e.g., ascites, variceal bleeding, or encephalopathy).
* Creatinine clearance less than 70 milliliter per minutes (mL/min).
* Alanine aminotransferase >10 times ULN at screening or history of acute exacerbation leading to transient decompensation.
* Haemoglobin <8 grams per deciliter (g/dL), absolute neutrophil count <1.0 x 10^9 per Liter, platelets <75 x 10^9 per Liter.
* Documented co-infection with hepatitis A (HAV), hepatitis C (HCV), hepatitis delta virus (HDV), hepatitis E virus (HEV) or Human immunodeficiency virus (HIV). For HCV co-infection, subjects who are anti-HCV positive and in whom HCV RNA is undetectable are considered to be not eligible for enrolment.
* Evidence of active liver disease due to autoimmune hepatitis (antinuclear antibody titre >1:160)
* Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the Investigator, would interfere with subject treatment, assessment or compliance with the protocol. This would include any uncontrolled clinically significant renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders, pathological fractures or cancer.
* Active alcohol or drug abuse or history of alcohol or drug abuse considered by the Investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results.
* A female who is breastfeeding or plan to breast.
* Use of immunosuppressive therapy, immunomodulatory therapy [including Pegylated interferon (PEG-IFN) and short-acting interferon or thymosin alpha], systemic cytotoxic agents within the previous 6 months prior to screening.
* Planned for liver transplantation or previous liver transplantation.
* Receipt of TDF within 6 months prior to screening.
* Therapy with nephrotoxic drugs (e.g., aminoglycosides, amphotercin B, vancomycin, cidofovir, foscarnet, cis-platinum, pentamidine etc.) or competitors of renal excretion (e.g., probenecid) within 2 months prior to study screening or the expectation that subject will receive any of these during the course of the study.
* History of hypersensitivity to nucleoside and/or nucleotide analogues and/or any component of study medication.
* Inability to comply with study requirements as determined by the study Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- China (7):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted to evaluate the efficacy and safety of Tenofovir Disoproxil Fumarate treatment in Chinese chronic hepatitis B (CHB) participants following failure of multiple Nucleos(t)ide analogues(NAs) at different centers in China.
Pre-assignment Details: A total of 281 participants were screened; of these 68 were screen failures. A total of 213 participants entered the treatment phase of the study.
Groups:
- Tenofovir Disoproxil Fumerate 300 mg: Participants received an open-label treatment of Tenofovir Disoproxil Fumarate 300 mg orally once daily for 144-weeks.
Period: Overall Study
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Started | 213
Completed | 204
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 4
Not completed — Pregnancy | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 186
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 213

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) <20 International Unit Per Milliliter (IU/mL) at Week 144
Description: HBV DNA level were analyzed using the sensitive HBV test in central laboratory using Roche cobas Taqman HBV test from the blood samples collected at Week 144. A 95 percent confidence interval (CI) was constructed by normal approximation and continuity correction method. Percentage of participants with serum HBV DNA <20 IU/mL at Week 144 have been presented. The Modified Intent-to-treat (mITT) Population was defined as all recruited participants who received at least one dose of study medication.
Time Frame: At Week 144
Population: mITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 213
Percentage of Participants | 77.0

2. Secondary Outcome: Percentage of Participants With Serum HBV DNA <20 IU/mL and Serum HBV DNA <69 IU/mL at Weeks 48 and 96
Description: HBV DNA level were analyzed using the sensitive HBV test in central laboratory using Roche cobas Taqman HBV test from the blood samples collected at Weeks 48 and 96. Virological response was assessed by proportion of participants with serum serum HBV <20 IU/mL and <69 IU/mL at Weeks 48 and 96. Percentage of participants with serum HBV DNA <20 IU/mL and <69 IU/mL at Weeks 48 and 96 have been presented.
Time Frame: At Weeks 48 and 96
Population: mITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 213
Percentage of Participants
  Week 48, HBV DNA <20 IU/mL | 46.9
  Week 48, HBV DNA <69 IU/mL | 76.5
  Week 96, HBV DNA <20 IU/mL | 61.0
  Week 96, HBV DNA <69 IU/mL | 84.0

3. Secondary Outcome: Percentage of Participants in the Subgroup With Confirmed Multi-drug Resistance Mutations at Baseline With Serum HBV DNA <20 IU/mL and Serum HBV DNA <69 IU/mL at Weeks 48, 96 and 144
Description: Serum samples were collected and analyzed for HBV DNA levels at indicated time points. Resistance surveillance of the HBV polymerase gene were performed by direct sequencing for all participants at Baseline. Day 0 was considered as Baseline. Percentage of participants in the subgroup with confirmed multi-drug resistance mutations at Baseline with serum HBV DNA <20 IU/mL and serum HBV DNA <69 IU/mL at Weeks 48, 96 and 144 have been presented.
Time Frame: At Weeks 48, 96, and 144
Population: mITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 213
Percentage of Participants
  Week 48, HBV DNA <20 IU/mL | 34.2
  Week 48, HBV DNA <69 IU/mL | 60.5
  Week 96, HBV DNA <20 IU/mL | 55.3
  Week 96, HBV DNA <69 IU/mL | 76.3
  Week 144, HBV DNA <20 IU/mL | 65.8
  Week 144, HBV DNA <69 IU/mL | 84.2

4. Secondary Outcome: Change From Baseline in Logarithm to the Base 10 (Log 10) Reduction in Serum HBV DNA at Week 48, 96 and 144
Description: Log10 reduction in serum HBV DNA was analyzed by patterns of mutation. The patterns of mutation were summarized by 2 categories. Category 1 included wild-type, LAM-R (Lamivudine-resistant), ADV-R (Adefovir-resistant) and ETV-R (Entecavir-resistant). Category 2 included Wild type, ADV-R single mutation, ADV-R double mutation and other mutation. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks 48,96, and 144
Population: mITT Population. All the participants in the study were analyzed (213 Participants) but only the participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Log 10 (IU/mL)
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 213
Log 10 (IU/mL)
  Category 1, Week 48, Wild type, n=57: number analyzed (Participants) | 57
  Category 1, Week 48, Wild type, n=57 | -2.2 (1.63)
  Category 1,Week 96, Wild type, n=57: number analyzed (Participants) | 57
  Category 1,Week 96, Wild type, n=57 | -2.3 (1.61)
  Category 1,Week 144, Wild type, n=56: number analyzed (Participants) | 56
  Category 1,Week 144, Wild type, n=56 | -2.4 (1.54)
  Category 1,Week 48, ADV-R, n=38: number analyzed (Participants) | 38
  Category 1,Week 48, ADV-R, n=38 | -3.0 (1.58)
  Category 1, Week 96, ADV-R, n=38: number analyzed (Participants) | 38
  Category 1, Week 96, ADV-R, n=38 | -3.3 (1.53)
  Category 1, Week 144, ADV-R, n=38: number analyzed (Participants) | 38
  Category 1, Week 144, ADV-R, n=38 | -3.5 (1.55)
  Category 1, Week 48, ETV-R, n=32: number analyzed (Participants) | 32
  Category 1, Week 48, ETV-R, n=32 | -3.2 (1.49)
  Category 1, Week 96, ETV-R, n=32: number analyzed (Participants) | 32
  Category 1, Week 96, ETV-R, n=32 | -3.4 (1.49)
  Category 1, Week 144, ETV-R, n=31: number analyzed (Participants) | 31
  Category 1, Week 144, ETV-R, n=31 | -3.6 (1.47)
  Category 1, Week 48, LAM-R, n=93: number analyzed (Participants) | 93
  Category 1, Week 48, LAM-R, n=93 | -3.1 (1.50)
  Category 1, Week 96, LAM-R, n=92: number analyzed (Participants) | 92
  Category 1, Week 96, LAM-R, n=92 | -3.3 (1.59)
  Category 1, Week 144,LAM-R, n=91: number analyzed (Participants) | 91
  Category 1, Week 144,LAM-R, n=91 | -3.2 (1.75)
  Category 2, Week 48, Wild type, n=57: number analyzed (Participants) | 57
  Category 2, Week 48, Wild type, n=57 | -2.2 (1.63)
  Category 2,Week 96, Wild type, n=57: number analyzed (Participants) | 57
  Category 2,Week 96, Wild type, n=57 | -2.3 (1.61)
  Category 2 Week 144, Wild type, n=56: number analyzed (Participants) | 56
  Category 2 Week 144, Wild type, n=56 | -2.4 (1.54)
  Category 2, Week 48, ADV-R single mutation, n=28: number analyzed (Participants) | 28
  Category 2, Week 48, ADV-R single mutation, n=28 | -2.9 (1.69)
  Category 2, Week 96, ADV-R, single mutation, n=28: number analyzed (Participants) | 28
  Category 2, Week 96, ADV-R, single mutation, n=28 | -3.3 (1.65)
  Category 2, Week 144, ADV-R single mutation, n=28: number analyzed (Participants) | 28
  Category 2, Week 144, ADV-R single mutation, n=28 | -3.5 (1.64)
  Category 2, Week 48,ADV-R double mutation, n=10: number analyzed (Participants) | 10
  Category 2, Week 48,ADV-R double mutation, n=10 | -3.2 (1.26)
  Category 2, Week 96, ADV-R double mutation, n=10: number analyzed (Participants) | 10
  Category 2, Week 96, ADV-R double mutation, n=10 | -3.3 (1.22)
  Category 1, Week 144, ADV-R double mutation, n=10: number analyzed (Participants) | 10
  Category 1, Week 144, ADV-R double mutation, n=10 | -3.5 (1.36)
  Category 2, Week 48, other mutation, n=113: number analyzed (Participants) | 113
  Category 2, Week 48, other mutation, n=113 | -3.1 (1.48)
  Category 2, Week 96, other mutation, n=112: number analyzed (Participants) | 112
  Category 2, Week 96, other mutation, n=112 | -3.2 (1.53)
  Category 2, Week 144, other mutation, n=110: number analyzed (Participants) | 110
  Category 2, Week 144, other mutation, n=110 | -3.2 (1.67)

5. Secondary Outcome: Percentage of Hepatitis B e Antigen (HBeAg) Positive Participants Achieving HBeAg Loss, HBeAg Seroconversion or Hepatitis B s Antigen (HBsAg) Loss and HBsAg Seroconversion at Weeks 48, 96, and 144
Description: Serological response was assessed at Weeks 48, 96 and 144 in participants with Positive HBeAg at Baseline (Day 0). It was presented as HBeAg Loss, HBeAg Seroconversion, HBsAg Loss and HBsAg Seroconversion. HBeAg Loss was defined as HBeAg changed to be negative. HBeAg seroconversion was defined as HBeAg changed to negative and HBeAb was positive. HBsAg Loss was defined as HBsAg changed to be negative. HBsAg seroconversion was defined as HBsAg changed to negative and HBsAb was positive.
Time Frame: At Weeks 48, 96 and 144
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 190
Percentage of Participants
  Week 48, HBeAg loss | 5.3
  Week 48, HBeAg seroconversion | 2.6
  Week 48, HBsAg loss | 0.5
  Week 48, HBsAg seroconversion | 0
  Week 96, HBeAg loss | 10.0
  Week 96, HBeAg seroconversion | 2.6
  Week 96, HBsAg loss | 0.5
  Week 96, HBsAg seroconversion | 0.5
  Week 144, HBeAg loss | 15.3
  Week 144, HBeAg seroconversion | 4.7
  Week 144, HBsAg loss | 1.1
  Week 144, HBsAg seroconversion | 0.5

6. Secondary Outcome: Percentage of HBeAg Negative Participants Achieving HBsAg Loss and HBsAg Seroconversion at Weeks 48, 96, and 144
Description: Serological response was assessed at Weeks 48, 96 and 144 in participants with negative HBeAg at Baseline (Day 0). HBsAg Loss was defined as HBsAg changed to be negative. HBsAg seroconversion was defined as HBsAg changed to negative and HBsAb was positive.
Time Frame: At Weeks 48,96, and 144
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 23
Percentage of Participants
  Week 48, HBsAg loss | 0
  Week 48, HBsAg seroconversion | 0
  Week 96, HBsAg loss | 0
  Week 96, HBsAg seroconversion | 0
  Week 144, HBsAg loss | 0
  Week 144, HBsAg seroconversion | 0

7. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Weeks 48, 96, and 144 in Participants Who Had Abnormal ALT at Baseline
Description: Blood samples were collected for evaluation of ALT at indicated time points. ALT normalization was defined as measurement less than or equal to the upper limit of the normal range. Normal range for ALT is 7 to 56 International Units per liter. Percentage of participants with ALT normalization at Weeks 48, 96, and 144 in Participants who had abnormal ALT at Baseline (Day 0) have been presented.
Time Frame: At Weeks 48, 96, and 144
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 61
Percentage of Participants
  Week 48 | 52.5
  Week 96 | 60.7
  Week 144 | 68.3

8. Secondary Outcome: Percentage of Participants Who Experienced Viral Breakthrough up to Week 144
Description: Viral breakthrough was defined as 1 log increase in HBV DNA from nadir determined by two sequential HBV DNA measurements. Percentage of participants who experienced viral breakthrough at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132 and 144 have been presented.
Time Frame: At Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120,132, and 144
Population: mITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 213
Percentage of Participants
  Week 24 | 0.5
  Week 36 | 0
  Week 48 | 0.5
  Week 60 | 0
  Week 72 | 0
  Week 84 | 0
  Week 96 | 0
  Week 108 | 0.5
  Week 120 | 0
  Week 132 | 0
  Week 144 | 0

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Non-serious TEAEs
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is defined as AE occurred on or after the first dose date of study drug, SAE is any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement or events associated with liver injury and impaired liver function. The Safety analysis (SA) Population was defined as all participants who received at least one dose of study medication and have at least one post Baseline safety assessment.
Time Frame: Up to Week 144
Population: Safety Analysis Population.
Measure: Number; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 213
Participants
  Any TEAEs | 124
  Serious TEAEs | 20
  Non-serious TEAEs | 117

10. Secondary Outcome: Change From Baseline in Hematology Parameters: White Blood Cells (WBC), Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Blood samples were collected to analyze the hematology parameters: WBC, basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelets. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks 24, 48, 72, 96, 120 and 144
Population: Safety analysis Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Billion cells per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 208
Billion cells per liter
  Week 24, WBC, n=208 | 0.19 (1.409)
  Week 48, WBC, n=208 | 0.15 (1.470)
  Week 72, WBC, n=207: number analyzed (Participants) | 207
  Week 72, WBC, n=207 | 0.13 (1.553)
  Week 96, WBC, n=207: number analyzed (Participants) | 207
  Week 96, WBC, n=207 | 0.07 (1.504)
  Week 120, WBC, n=204: number analyzed (Participants) | 204
  Week 120, WBC, n=204 | 0.10 (1.566)
  Week 144, WBC, n=204: number analyzed (Participants) | 204
  Week 144, WBC, n=204 | 0.12 (1.484)
  Week 24, Neutrophils, n=208 | 0.15 (1.322)
  Week 48, Neutrophils, n=208 | 0.09 (1.419)
  Week 72, Neutrophils, n=207: number analyzed (Participants) | 207
  Week 72, Neutrophils, n=207 | 0.10 (1.388)
  Week 96, Neutrophils, n=207: number analyzed (Participants) | 207
  Week 96, Neutrophils, n=207 | 0.05 (1.414)
  Week 120, Neutrophils, n=204: number analyzed (Participants) | 204
  Week 120, Neutrophils, n=204 | 0.14 (1.400)
  Week 144, Neutrophils, n=204: number analyzed (Participants) | 204
  Week 144, Neutrophils, n=204 | 0.12 (1.293)
  Week 24, Lymphocytes, n=208 | 0.02 (0.390)
  Week 48, Lymphocytes, n=208 | 0.05 (0.396)
  Week 72, Lymphocytes, n=207: number analyzed (Participants) | 207
  Week 72, Lymphocytes, n=207 | 0.02 (0.490)
  Week 96, Lymphocytes, n=207: number analyzed (Participants) | 207
  Week 96, Lymphocytes, n=207 | 0.02 (0.439)
  Week 120, Lymphocytes, n=204: number analyzed (Participants) | 204
  Week 120, Lymphocytes, n=204 | -0.05 (0.459)
  Week 144, Lymphocyte, n=204: number analyzed (Participants) | 204
  Week 144, Lymphocyte, n=204 | 0.00 (0.443)
  Week 24, Monocytes, n=208 | -0.001 (0.1069)
  Week 48, Monocytes, n=208 | 0.004 (0.1163)
  Week 72, Monocytes, n=207: number analyzed (Participants) | 207
  Week 72, Monocytes, n=207 | -0.010 (0.1177)
  Week 96, Monocytes, n=207: number analyzed (Participants) | 207
  Week 96, Monocytes, n=207 | -0.009 (0.1123)
  Week 120, Monocytes, n=204: number analyzed (Participants) | 204
  Week 120, Monocytes, n=204 | -0.006 (0.1209)
  Week 144, Monocytes, n=204: number analyzed (Participants) | 204
  Week 144, Monocytes, n=204 | -0.008 (0.1285)
  Week 24, Eosinophils, n=208 | 0.02 (0.153)
  Week 48, Eosinophils, n=208 | -0.00 (0.079)
  Week 72, Eosinophils, n=207: number analyzed (Participants) | 207
  Week 72, Eosinophils, n=207 | 0.02 (0.225)
  Week 96, Eosinophils, n=207: number analyzed (Participants) | 207
  Week 96, Eosinophils, n=207 | -0.00 (0.076)
  Week 120, Eosinophils, n=204: number analyzed (Participants) | 204
  Week 120, Eosinophils, n=204 | 0.00 (0.092)
  Week 144, Eosinophils, n=204: number analyzed (Participants) | 204
  Week 144, Eosinophils, n=204 | 0.00 (0.097)
  Week 24, Basophils, n=208 | 0.00 (0.027)
  Week 48, Basophils, n=208 | 0.00 (0.023)
  Week 72, Basophils, n=207: number analyzed (Participants) | 207
  Week 72, Basophils, n=207 | -0.00 (0.025)
  Week 96, Basophils, n=207: number analyzed (Participants) | 207
  Week 96, Basophils, n=207 | -0.00 (0.024)
  Week 120, Basophils, n=203: number analyzed (Participants) | 203
  Week 120, Basophils, n=203 | 0.00 (0.025)
  Week 144, Basophils, n=203: number analyzed (Participants) | 203
  Week 144, Basophils, n=203 | 0.00 (0.025)
  Week 24, Platelets, n=208 | 3.5 (27.07)
  Week 48, Platelets, n=208 | 2.5 (29.38)
  Week 72, Platelets, n=207: number analyzed (Participants) | 207
  Week 72, Platelets, n=207 | 1.9 (33.74)
  Week 96, Platelets, n=207: number analyzed (Participants) | 207
  Week 96, Platelets, n=207 | 3.9 (33.20)
  Week 120, Platelets, n=204: number analyzed (Participants) | 204
  Week 120, Platelets, n=204 | 7.2 (33.48)
  Week 144, Platelets, n=204: number analyzed (Participants) | 204
  Week 144, Platelets, n=204 | 9.3 (34.74)

11. Secondary Outcome: Change From Baseline in Hemoglobin (Hb)
Description: Blood samples were collected to analyze Hb values. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks 24, 48, 72, 96, 120 and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 208
Grams per liter
  Week 24, n=208 | 2.4 (6.53)
  Week 48, n=208 | -0.2 (7.04)
  Week 72, n=207: number analyzed (Participants) | 207
  Week 72, n=207 | -0.2 (7.68)
  Week 96, n=207: number analyzed (Participants) | 207
  Week 96, n=207 | -1.0 (8.67)
  Week 120, n=204: number analyzed (Participants) | 204
  Week 120, n=204 | -1.0 (8.86)
  Week 144, n=204: number analyzed (Participants) | 204
  Week 144, n=204 | -0.2 (9.24)

12. Secondary Outcome: Change From Baseline in Red Blood Cells (RBC)
Description: Blood samples were collected to analyze RBC values. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks 24, 48, 72, 96, 120 and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 208
Trillion cells per liter
  Week 24, n=208 | 0.13 (0.254)
  Week 48, n=208 | 0.05 (0.259)
  Week 72, n=207: number analyzed (Participants) | 207
  Week 72, n=207 | 0.07 (0.268)
  Week 96, n=207: number analyzed (Participants) | 207
  Week 96, n=207 | 0.02 (0.294)
  Week 120, n=204: number analyzed (Participants) | 204
  Week 120, n=204 | 0.08 (0.291)
  Week 144, n=204: number analyzed (Participants) | 204
  Week 144, n=204 | 0.06 (0.305)

13. Secondary Outcome: Change From Baseline in Chemistry Parameters: ALT, Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-Glutamyltransferase (GGT), Creatinine Phosphokinase (CK), Lactose Dehydrogenase (LDH)
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP, AST, GGT, CK, LDH. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks 12,24,36,48,60,72,84,96,108,120,132,and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 209
International units per liter
  Week 12, ALT, n=209 | 1.66 (54.582)
  Week 24, ALT, n=208: number analyzed (Participants) | 208
  Week 24, ALT, n=208 | -2.80 (51.195)
  Week 36, ALT, n=209 | -4.57 (51.811)
  Week 48, ALT, n=208: number analyzed (Participants) | 208
  Week 48, ALT, n=208 | -7.07 (50.986)
  Week 60, ALT, n=208: number analyzed (Participants) | 208
  Week 60, ALT, n=208 | -9.20 (50.312)
  Week 72, ALT, n=207: number analyzed (Participants) | 207
  Week 72, ALT, n=207 | -8.12 (51.538)
  Week 84, ALT, n=207: number analyzed (Participants) | 207
  Week 84, ALT, n=207 | -10.53 (51.781)
  Week 96, ALT, n=207: number analyzed (Participants) | 207
  Week 96, ALT, n=207 | -9.13 (54.323)
  Week 108, ALT, n=205: number analyzed (Participants) | 205
  Week 108, ALT, n=205 | -11.25 (52.277)
  Week 120, ALT, n=205: number analyzed (Participants) | 205
  Week 120, ALT, n=205 | -11.95 (51.584)
  Week 132, ALT, n=205: number analyzed (Participants) | 205
  Week 132, ALT, n=205 | -11.56 (51.594)
  Week 144, ALT, n=204: number analyzed (Participants) | 204
  Week 144, ALT, n=204 | -10.97 (53.326)
  Week 12, AST, n=209 | -1.68 (44.258)
  Week 24, AST, n=208: number analyzed (Participants) | 208
  Week 24, AST, n=208 | -3.20 (44.506)
  Week 36, AST, n=209 | -2.93 (45.755)
  Week 48, AST, n=205: number analyzed (Participants) | 205
  Week 48, AST, n=205 | -4.23 (45.393)
  Week 60, AST, n=208: number analyzed (Participants) | 208
  Week 60, AST, n=208 | -4.68 (44.969)
  Week 72, AST, n=207: number analyzed (Participants) | 207
  Week 72, AST, n=207 | -4.43 (44.901)
  Week 84, AST, n=207: number analyzed (Participants) | 207
  Week 84, AST, n=207 | -5.56 (45.435)
  Week 96, AST, n=207: number analyzed (Participants) | 207
  Week 96, AST, n=207 | -4.37 (46.008)
  Week 108, AST, n=205: number analyzed (Participants) | 205
  Week 108, AST, n=205 | -5.81 (45.818)
  Week 120, AST, n=205: number analyzed (Participants) | 205
  Week 120, AST, n=205 | -5.67 (45.645)
  Week 132, AST, n=205: number analyzed (Participants) | 205
  Week 132, AST, n=205 | -6.05 (45.290)
  Week 144, AST, n=204: number analyzed (Participants) | 204
  Week 144, AST, n=204 | -5.85 (46.176)
  Week 12, ALP, n=208: number analyzed (Participants) | 208
  Week 12, ALP, n=208 | 4.46 (11.718)
  Week 24, ALP, n=208: number analyzed (Participants) | 208
  Week 24, ALP, n=208 | 7.22 (13.819)
  Week 36, ALP, n=209 | 6.27 (12.609)
  Week 48, ALP, n=208: number analyzed (Participants) | 208
  Week 48, ALP, n=208 | 8.24 (12.225)
  Week 60, ALP, n=208: number analyzed (Participants) | 208
  Week 60, ALP, n=208 | 8.75 (14.321)
  Week 72, ALP, n=207: number analyzed (Participants) | 207
  Week 72, ALP, n=207 | 10.06 (16.259)
  Week 84, ALP, n=207: number analyzed (Participants) | 207
  Week 84, ALP, n=207 | 7.32 (14.478)
  Week 96, ALP, n=207: number analyzed (Participants) | 207
  Week 96, ALP, n=207 | 8.73 (13.854)
  Week 108, ALP, n=205: number analyzed (Participants) | 205
  Week 108, ALP, n=205 | 7.62 (15.102)
  Week 120, ALP, n=205: number analyzed (Participants) | 205
  Week 120, ALP, n=205 | 7.54 (17.844)
  Week 132, ALP, n=205: number analyzed (Participants) | 205
  Week 132, ALP, n=205 | 7.36 (15.802)
  Week 144, ALP, n=205: number analyzed (Participants) | 205
  Week 144, ALP, n=205 | 7.14 (15.099)
  Week 12, GGT, n=208: number analyzed (Participants) | 208
  Week 12, GGT, n=208 | -1.83 (18.966)
  Week 24, GGT, n=208: number analyzed (Participants) | 208
  Week 24, GGT, n=208 | -1.83 (19.853)
  Week 36, GGT, n=209 | -2.25 (20.205)
  Week 48, GGT, n=207: number analyzed (Participants) | 207
  Week 48, GGT, n=207 | -1.90 (20.760)
  Week 60, GGT, n=208: number analyzed (Participants) | 208
  Week 60, GGT, n=208 | -1.25 (22.512)
  Week 72, GGT, n=207: number analyzed (Participants) | 207
  Week 72, GGT, n=207 | -1.45 (23.700)
  Week 84, GGT, n=207: number analyzed (Participants) | 207
  Week 84, GGT, n=207 | -2.10 (21.532)
  Week 96, GGT, n=207: number analyzed (Participants) | 207
  Week 96, GGT, n=207 | -2.50 (21.436)
  Week 108, GGT, n=205: number analyzed (Participants) | 205
  Week 108, GGT, n=205 | -1.62 (22.053)
  Week 120, GGT, n=205: number analyzed (Participants) | 205
  Week 120, GGT, n=205 | -1.61 (22.872)
  Week 132, GGT, n=205: number analyzed (Participants) | 205
  Week 132, GGT, n=205 | -1.80 (21.897)
  Week 144, GGT, n=203: number analyzed (Participants) | 203
  Week 144, GGT, n=203 | -0.76 (25.363)
  Week 12, CK, n=206: number analyzed (Participants) | 206
  Week 12, CK, n=206 | 10.84 (525.680)
  Week 24, CK, n=198: number analyzed (Participants) | 198
  Week 24, CK, n=198 | -9.28 (108.221)
  Week 36, CK, n=201: number analyzed (Participants) | 201
  Week 36, CK, n=201 | 13.87 (315.156)
  Week 48 CK, n=206: number analyzed (Participants) | 206
  Week 48 CK, n=206 | -21.58 (202.083)
  Week 60, CK, n=205: number analyzed (Participants) | 205
  Week 60, CK, n=205 | -22.26 (207.666)
  Week 72, CK, n=206: number analyzed (Participants) | 206
  Week 72, CK, n=206 | -13.45 (209.963)
  Week 84, CK, n=207: number analyzed (Participants) | 207
  Week 84, CK, n=207 | -17.40 (204.800)
  Week 96, CK, n=207: number analyzed (Participants) | 207
  Week 96, CK, n=207 | 26.58 (415.775)
  Week 108, CK, n=199: number analyzed (Participants) | 199
  Week 108, CK, n=199 | -20.58 (211.398)
  Week 120, CK, n=203: number analyzed (Participants) | 203
  Week 120, CK, n=203 | 0.59 (261.655)
  Week 132, CK, n=204: number analyzed (Participants) | 204
  Week 132, CK, n=204 | -19.34 (214.775)
  Week 144, CK, n=204: number analyzed (Participants) | 204
  Week 144, CK, n=204 | -7.17 (270.074)
  Week 12, LDH, n=209 | 1.66 (54.582)
  Week 24, LDH, n=208: number analyzed (Participants) | 208
  Week 24, LDH, n=208 | -2.80 (51.195)
  Week 36, LDH, n=209 | -4.57 (51.811)
  Week 48, LDH, n=208: number analyzed (Participants) | 208
  Week 48, LDH, n=208 | -7.07 (50.986)
  Week 60, LDH, n=208: number analyzed (Participants) | 208
  Week 60, LDH, n=208 | -9.20 (50.312)
  Week 72, LDH, n=207: number analyzed (Participants) | 207
  Week 72, LDH, n=207 | -8.12 (51.538)
  Week 84, LDH, n=207: number analyzed (Participants) | 207
  Week 84, LDH, n=207 | -10.53 (51.781)
  Week 96, LDH, n=207: number analyzed (Participants) | 207
  Week 96, LDH, n=207 | -9.13 (54.323)
  Week 108, LDH, n=205: number analyzed (Participants) | 205
  Week 108, LDH, n=205 | -11.25 (52.277)
  Week 120, LDH, n=205: number analyzed (Participants) | 205
  Week 120, LDH, n=205 | -11.95 (51.584)
  Week 132, LDH, n=205: number analyzed (Participants) | 205
  Week 132, LDH, n=205 | -11.56 (51.594)
  Week 144, LDH, n=204: number analyzed (Participants) | 204
  Week 144, LDH, n=204 | -10.97 (53.326)

14. Secondary Outcome: Change From Baseline in Chemistry Parameters: Total Billirubin, Direct Bilirubin, Serum Creatinine
Description: Blood samples were collected to analyze the chemistry parameters: total billirubin,direct bilirubin and serum creatinine. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks, 12,24,36,48,60,72,84,96,108,120,132,and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 209
Micromoles per liter
  Week 12, total bilirubin, n=209 | -0.506 (4.8201)
  Week 24, total bilirubin, n=208: number analyzed (Participants) | 208
  Week 24, total bilirubin, n=208 | -0.755 (5.0494)
  Week 36, total bilirubin, n=209 | -0.878 (5.0063)
  Week 48, total bilirubin, n=207: number analyzed (Participants) | 207
  Week 48, total bilirubin, n=207 | -0.167 (4.8371)
  Week 60, total bilirubin, n=208: number analyzed (Participants) | 208
  Week 60, total bilirubin, n=208 | -0.334 (4.9175)
  Week 72, total bilirubin, n=207: number analyzed (Participants) | 207
  Week 72, total bilirubin, n=207 | -1.209 (5.1706)
  Week 84, total bilirubin, n=207: number analyzed (Participants) | 207
  Week 84, total bilirubin, n=207 | -1.112 (5.0813)
  Week 96, total bilirubin, n=207: number analyzed (Participants) | 207
  Week 96, total bilirubin, n=207 | -0.780 (5.1218)
  Week 108, total bilirubin, n=205: number analyzed (Participants) | 205
  Week 108, total bilirubin, n=205 | -0.795 (5.7857)
  Week 120, total bilirubin, n=205: number analyzed (Participants) | 205
  Week 120, total bilirubin, n=205 | -1.021 (5.3998)
  Week 132, total bilirubin, n=205: number analyzed (Participants) | 205
  Week 132, total bilirubin, n=205 | -1.471 (4.8998)
  Week 144, total bilirubin, n=204: number analyzed (Participants) | 204
  Week 144, total bilirubin, n=204 | -0.869 (5.4163)
  Week 12, direct bilirubin, n=209 | -0.181 (2.6421)
  Week 24, direct bilirubin, n=208: number analyzed (Participants) | 208
  Week 24, direct bilirubin, n=208 | -0.360 (2.2236)
  Week 36, direct bilirubin, n=208: number analyzed (Participants) | 208
  Week 36, direct bilirubin, n=208 | -0.541 (3.2564)
  Week 48, direct bilirubin, n=207: number analyzed (Participants) | 207
  Week 48, direct bilirubin, n=207 | -0.085 (3.0478)
  Week 60, direct bilirubin, n=208: number analyzed (Participants) | 208
  Week 60, direct bilirubin, n=208 | -0.111 (3.1364)
  Week 72, direct bilirubin, n=207: number analyzed (Participants) | 207
  Week 72, direct bilirubin, n=207 | -0.654 (3.7846)
  Week 84, direct bilirubin, n=207: number analyzed (Participants) | 207
  Week 84, direct bilirubin, n=207 | -0.797 (3.6592)
  Week 96, direct bilirubin, n=207: number analyzed (Participants) | 207
  Week 96, direct bilirubin, n=207 | -0.711 (3.3849)
  Week 108, direct bilirubin, n=205: number analyzed (Participants) | 205
  Week 108, direct bilirubin, n=205 | -0.632 (3.4657)
  Week 120, direct bilirubin, n=205: number analyzed (Participants) | 205
  Week 120, direct bilirubin, n=205 | -0.802 (3.6175)
  Week 132, direct bilirubin, n=205: number analyzed (Participants) | 205
  Week 132, direct bilirubin, n=205 | -0.805 (3.1588)
  Week 144, direct bilirubin, n=204: number analyzed (Participants) | 204
  Week 144, direct bilirubin, n=204 | -0.573 (2.8964)
  Week 12, serum creatinine, n=209 | 2.94 (7.089)
  Week 24, serum creatinine, n=208: number analyzed (Participants) | 208
  Week 24, serum creatinine, n=208 | 1.16 (6.934)
  Week 36, serum creatinine, n=209 | 0.67 (7.743)
  Week 48, serum creatinine, n=208: number analyzed (Participants) | 208
  Week 48, serum creatinine, n=208 | 1.43 (7.480)
  Week 60, serum creatinine, n=208: number analyzed (Participants) | 208
  Week 60, serum creatinine, n=208 | 0.25 (8.181)
  Week 72, serum creatinine, n=206: number analyzed (Participants) | 206
  Week 72, serum creatinine, n=206 | -1.00 (7.583)
  Week 84, serum creatinine, n=207: number analyzed (Participants) | 207
  Week 84, serum creatinine, n=207 | -0.65 (9.075)
  Week 96, serum creatinine, n=207: number analyzed (Participants) | 207
  Week 96, serum creatinine, n=207 | 0.22 (9.013)
  Week 108, serum creatinine, n=204: number analyzed (Participants) | 204
  Week 108, serum creatinine, n=204 | -0.28 (8.511)
  Week 120, serum creatinine, n=205: number analyzed (Participants) | 205
  Week 120, serum creatinine, n=205 | -1.22 (8.844)
  Week 132, serum creatinine, n=205: number analyzed (Participants) | 205
  Week 132, serum creatinine, n=205 | -0.81 (8.250)
  Week 144, serum creatinine, n=203: number analyzed (Participants) | 203
  Week 144, serum creatinine, n=203 | -1.28 (8.610)

15. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin, Total Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin and total protein. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks, 12,24,36,48,60,72,84,96,108,120,132,and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 209
Grams per liter
  Week 12, albumin, n=209 | 0.22 (2.766)
  Week 24, albumin, n=208: number analyzed (Participants) | 208
  Week 24, albumin, n=208 | 0.54 (2.722)
  Week 36, albumin, n=209 | 0.04 (2.545)
  Week 48, albumin, n=208: number analyzed (Participants) | 208
  Week 48, albumin, n=208 | 0.24 (2.687)
  Week 60, albumin, n=208: number analyzed (Participants) | 208
  Week 60, albumin, n=208 | 0.38 (2.757)
  Week 72, albumin, n=207: number analyzed (Participants) | 207
  Week 72, albumin, n=207 | 0.49 (2.890)
  Week 84, albumin, n=207: number analyzed (Participants) | 207
  Week 84, albumin, n=207 | -0.03 (3.021)
  Week 96, albumin, n=207: number analyzed (Participants) | 207
  Week 96, albumin, n=207 | 0.13 (2.980)
  Week 108, albumin, n=205: number analyzed (Participants) | 205
  Week 108, albumin, n=205 | -0.56 (2.932)
  Week 120, albumin, n=205: number analyzed (Participants) | 205
  Week 120, albumin, n=205 | 0.17 (3.272)
  Week 132, albumin, n=205: number analyzed (Participants) | 205
  Week 132, albumin, n=205 | 0.51 (2.942)
  Week 144, albumin, n=204: number analyzed (Participants) | 204
  Week 144, albumin, n=204 | 0.48 (3.171)
  Week 12, total protein, n=209 | 0.31 (4.220)
  Week 24, total protein, n=207: number analyzed (Participants) | 207
  Week 24, total protein, n=207 | 0.92 (4.322)
  Week 36, total protein, n=209 | -0.30 (4.280)
  Week 48, total protein, n=208: number analyzed (Participants) | 208
  Week 48, total protein, n=208 | -0.53 (4.240)
  Week 60, total protein, n=208: number analyzed (Participants) | 208
  Week 60, total protein, n=208 | -0.32 (4.387)
  Week 72, total protein, n=207: number analyzed (Participants) | 207
  Week 72, total protein, n=207 | -0.26 (4.540)
  Week 84, total protein, n=207: number analyzed (Participants) | 207
  Week 84, total protein, n=207 | -0.57 (5.158)
  Week 96, total protein, n=207: number analyzed (Participants) | 207
  Week 96, total protein, n=207 | -0.44 (5.240)
  Week 108, total protein, n=205: number analyzed (Participants) | 205
  Week 108, total protein, n=205 | -0.21 (4.855)
  Week 120, total protein, n=205: number analyzed (Participants) | 205
  Week 120, total protein, n=205 | 0.95 (5.361)
  Week 132, total protein, n=205: number analyzed (Participants) | 205
  Week 132, total protein, n=205 | 1.00 (4.494)
  Week 144, total protein, n=204: number analyzed (Participants) | 204
  Week 144, total protein, n=204 | 0.94 (4.794)

16. Secondary Outcome: Change From Baseline in Chemistry Parameter: Blood Urea Nitrogen (BUN), Potassium, Sodium, Chloridian, Phosphorus, Calcium and Fasting Blood Glucose.
Description: Blood samples were collected to analyze the chemistry parameters: BUN, potassium, sodium, chloridian, phosphorus, calcium and fasting blood glucose. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks, 12,24,36,48,60,72,84,96,108,120,132,and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 209
Millimoles per liter
  Week 12, BUN, n=209 | -0.020 (1.0496)
  Week 24, BUN, n=208: number analyzed (Participants) | 208
  Week 24, BUN, n=208 | 0.069 (1.0725)
  Week 36, BUN, n=209 | 0.081 (1.0921)
  Week 48, BUN, n=208: number analyzed (Participants) | 208
  Week 48, BUN, n=208 | 0.075 (1.0907)
  Week 60, BUN, n=208: number analyzed (Participants) | 208
  Week 60, BUN, n=208 | 0.078 (1.0372)
  Week 72, BUN, n=206: number analyzed (Participants) | 206
  Week 72, BUN, n=206 | 0.119 (1.1114)
  Week 84, BUN, n=207: number analyzed (Participants) | 207
  Week 84, BUN, n=207 | 0.164 (1.0819)
  Week 96, BUN, n=207: number analyzed (Participants) | 207
  Week 96, BUN, n=207 | 0.100 (1.0482)
  Week 108, BUN, n=204: number analyzed (Participants) | 204
  Week 108, BUN, n=204 | 0.051 (1.1279)
  Week 120, BUN, n=205: number analyzed (Participants) | 205
  Week 120, BUN, n=205 | 0.110 (1.1672)
  Week 132, BUN, n=205: number analyzed (Participants) | 205
  Week 132, BUN, n=205 | 0.090 (1.1443)
  Week 144, BUN, n=203: number analyzed (Participants) | 203
  Week 144, BUN, n=203 | 0.193 (1.2236)
  Week 12, Potassium, n=209 | -0.029 (0.3391)
  Week 24, Potassium, n=208: number analyzed (Participants) | 208
  Week 24, Potassium, n=208 | 0.028 (0.3659)
  Week 36, Potassium, n=209 | 0.073 (0.3681)
  Week 48, Potassium, n=208: number analyzed (Participants) | 208
  Week 48, Potassium, n=208 | 0.016 (0.3206)
  Week 60, Potassium, n=208: number analyzed (Participants) | 208
  Week 60, Potassium, n=208 | 0.014 (0.3622)
  Week 72, Potassium, n=206: number analyzed (Participants) | 206
  Week 72, Potassium, n=206 | -0.032 (0.3402)
  Week 84, Potassium, n=206: number analyzed (Participants) | 206
  Week 84, Potassium, n=206 | 0.022 (0.3617)
  Week 96, Potassium, n=206: number analyzed (Participants) | 206
  Week 96, Potassium, n=206 | -0.019 (0.3357)
  Week 108, Potassium, n=204: number analyzed (Participants) | 204
  Week 108, Potassium, n=204 | -0.023 (0.3326)
  Week 120, Potassium, n=204: number analyzed (Participants) | 204
  Week 120, Potassium, n=204 | -0.002 (0.3221)
  Week 132, Potassium, n=204: number analyzed (Participants) | 204
  Week 132, Potassium, n=204 | 0.001 (0.3531)
  Week 144, Potassium, n=204: number analyzed (Participants) | 204
  Week 144, Potassium, n=204 | -0.000 (0.3851)
  Week 12, Sodium, n=209 | 0.31 (2.227)
  Week 24, Sodium, n=208: number analyzed (Participants) | 208
  Week 24, Sodium, n=208 | 0.52 (2.514)
  Week 36, Sodium, n=209 | 0.23 (2.437)
  Week 48, Sodium, n=208: number analyzed (Participants) | 208
  Week 48, Sodium, n=208 | 0.40 (2.781)
  Week 60, Sodium, n=208: number analyzed (Participants) | 208
  Week 60, Sodium, n=208 | 0.59 (2.569)
  Week 72, Sodium, n=206: number analyzed (Participants) | 206
  Week 72, Sodium, n=206 | 0.47 (2.631)
  Week 84, Sodium, n=207: number analyzed (Participants) | 207
  Week 84, Sodium, n=207 | 0.54 (2.689)
  Week 96, Sodium, n=206: number analyzed (Participants) | 206
  Week 96, Sodium, n=206 | 0.44 (2.388)
  Week 108, Sodium, n=204: number analyzed (Participants) | 204
  Week 108, Sodium, n=204 | 0.05 (2.352)
  Week 120, Sodium, n=204: number analyzed (Participants) | 204
  Week 120, Sodium, n=204 | 0.03 (3.332)
  Week 132, Sodium, n=204: number analyzed (Participants) | 204
  Week 132, Sodium, n=204 | 0.35 (2.672)
  Week 144, Sodium, n=204: number analyzed (Participants) | 204
  Week 144, Sodium, n=204 | 0.13 (2.642)
  Week 12, Chloridion n=209 | -0.23 (3.271)
  Week 24, Chloridion, n=208: number analyzed (Participants) | 208
  Week 24, Chloridion, n=208 | -0.32 (3.834)
  Week 36, Chloridion, n=209 | -0.50 (3.453)
  Week 48, Chloridion, n=208: number analyzed (Participants) | 208
  Week 48, Chloridion, n=208 | -0.31 (3.601)
  Week 60, Chloridion, n=208: number analyzed (Participants) | 208
  Week 60, Chloridion, n=208 | -0.37 (3.305)
  Week 72, Chloridion, n=206: number analyzed (Participants) | 206
  Week 72, Chloridion, n=206 | -0.30 (3.388)
  Week 84, Chloridion, n=207: number analyzed (Participants) | 207
  Week 84, Chloridion, n=207 | -0.38 (3.519)
  Week 96, Chloridion, n=206: number analyzed (Participants) | 206
  Week 96, Chloridion, n=206 | 0.04 (3.418)
  Week 108, Chloridion, n=204: number analyzed (Participants) | 204
  Week 108, Chloridion, n=204 | -0.27 (3.587)
  Week 120, Chloridion, n=204: number analyzed (Participants) | 204
  Week 120, Chloridion, n=204 | -0.17 (4.309)
  Week 132, Chloridion, n=204: number analyzed (Participants) | 204
  Week 132, Chloridion, n=204 | -0.14 (3.717)
  Week 144, Chloridion, n=204: number analyzed (Participants) | 204
  Week 144, Chloridion, n=204 | -0.28 (3.855)
  Week 12, Phosphorus, n=209 | -0.018 (0.1607)
  Week 24, Phosphorus, n=208: number analyzed (Participants) | 208
  Week 24, Phosphorus, n=208 | -0.001 (0.1662)
  Week 36, Phosphorus, n=209 | -0.001 (0.1779)
  Week 48, Phosphorus, n=208: number analyzed (Participants) | 208
  Week 48, Phosphorus, n=208 | -0.008 (0.1634)
  Week 60, Phosphorus, n=208: number analyzed (Participants) | 208
  Week 60, Phosphorus, n=208 | 0.004 (0.1685)
  Week 72, Phosphorus, n=207: number analyzed (Participants) | 207
  Week 72, Phosphorus, n=207 | -0.011 (0.1713)
  Week 84, Phosphorus, n=207: number analyzed (Participants) | 207
  Week 84, Phosphorus, n=207 | -0.023 (0.1736)
  Week 96, Phosphorus, n=206: number analyzed (Participants) | 206
  Week 96, Phosphorus, n=206 | -0.019 (0.1669)
  Week 108, Phosphorus, n=201: number analyzed (Participants) | 201
  Week 108, Phosphorus, n=201 | -0.008 (0.1779)
  Week 120, Phosphorus, n=203: number analyzed (Participants) | 203
  Week 120, Phosphorus, n=203 | -0.015 (0.1687)
  Week 132, Phosphorus, n=204: number analyzed (Participants) | 204
  Week 132, Phosphorus, n=204 | 0.002 (0.1757)
  Week 144, Phosphorus, n=204: number analyzed (Participants) | 204
  Week 144, Phosphorus, n=204 | -0.016 (0.1692)
  Week 12, Calcium, n=209 | -0.005 (0.1172)
  Week 24, Calcium, n=208: number analyzed (Participants) | 208
  Week 24, Calcium, n=208 | -0.027 (0.1289)
  Week 36, Calcium, n=209 | -0.030 (0.1432)
  Week 48, Calcium, n=208: number analyzed (Participants) | 208
  Week 48, Calcium, n=208 | -0.041 (0.1375)
  Week 60, Calcium, n=208: number analyzed (Participants) | 208
  Week 60, Calcium, n=208 | -0.038 (0.1365)
  Week 72, Calcium, n=207: number analyzed (Participants) | 207
  Week 72, Calcium, n=207 | -0.061 (0.1296)
  Week 84, Calcium, n=207: number analyzed (Participants) | 207
  Week 84, Calcium, n=207 | -0.060 (0.1321)
  Week 96, Calcium, n=206: number analyzed (Participants) | 206
  Week 96, Calcium, n=206 | -0.051 (0.1198)
  Week 108, Calcium, n=204: number analyzed (Participants) | 204
  Week 108, Calcium, n=204 | -0.062 (0.1290)
  Week 120, Calcium, n=204: number analyzed (Participants) | 204
  Week 120, Calcium, n=204 | -0.051 (0.1370)
  Week 132, Calcium, n=204: number analyzed (Participants) | 204
  Week 132, Calcium, n=204 | -0.052 (0.1235)
  Week 144, Calcium, n=204: number analyzed (Participants) | 204
  Week 144, Calcium, n=204 | -0.050 (0.1393)
  Week 12, Fasting blood glucose, n=205: number analyzed (Participants) | 205
  Week 12, Fasting blood glucose, n=205 | -0.088 (1.0006)
  Week 24, fasting blood glucose, n=208: number analyzed (Participants) | 208
  Week 24, fasting blood glucose, n=208 | -0.087 (0.8926)
  Week 36, fasting blood glucose, n=208: number analyzed (Participants) | 208
  Week 36, fasting blood glucose, n=208 | -0.150 (0.9535)
  Week 48, fasting blood glucose, n=208: number analyzed (Participants) | 208
  Week 48, fasting blood glucose, n=208 | -0.234 (0.8378)
  Week 60, fasting blood glucose, n=208: number analyzed (Participants) | 208
  Week 60, fasting blood glucose, n=208 | -0.206 (0.8658)
  Week 72, fasting blood glucose, n=202: number analyzed (Participants) | 202
  Week 72, fasting blood glucose, n=202 | -0.187 (0.8626)
  Week 84, fasting blood glucose, n=207: number analyzed (Participants) | 207
  Week 84, fasting blood glucose, n=207 | -0.143 (1.0564)
  Week 96, fasting blood glucose, n=206: number analyzed (Participants) | 206
  Week 96, fasting blood glucose, n=206 | -0.132 (1.1423)
  Week 108, fasting blood glucose, n=200: number analyzed (Participants) | 200
  Week 108, fasting blood glucose, n=200 | -0.230 (0.9042)
  Week 120, fasting blood glucose, n=204: number analyzed (Participants) | 204
  Week 120, fasting blood glucose, n=204 | -0.180 (0.9873)
  Week 132, fasting blood glucose, n=204: number analyzed (Participants) | 204
  Week 132, fasting blood glucose, n=204 | -0.151 (0.9312)
  Week 144, fasting blood glucose, n=204: number analyzed (Participants) | 204
  Week 144, fasting blood glucose, n=204 | -0.070 (1.0163)

17. Secondary Outcome: Change From Baseline in Chemistry Parameter: Creatinine Clearance Rate
Description: Blood samples were collected to analyze the chemistry parameter: creatinine clearance rate. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks, 12,24,36,48,60,72,84,96,108,120,132,and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Milliliter per minute
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 209
Milliliter per minute
  Week 12, n=208: number analyzed (Participants) | 208
  Week 12, n=208 | -4.564 (11.1192)
  Week 24, n=208: number analyzed (Participants) | 208
  Week 24, n=208 | -2.213 (11.2288)
  Week 36, n=209 | -2.311 (12.4693)
  Week 48, n=208: number analyzed (Participants) | 208
  Week 48, n=208 | -3.667 (12.3427)
  Week 60, n=208: number analyzed (Participants) | 208
  Week 60, n=208 | -2.053 (13.9768)
  Week 72, n=206: number analyzed (Participants) | 206
  Week 72, n=206 | -0.519 (13.1580)
  Week 84, n=207: number analyzed (Participants) | 207
  Week 84, n=207 | -1.065 (15.0315)
  Week 96, n=207: number analyzed (Participants) | 207
  Week 96, n=207 | -2.378 (13.8827)
  Week 108, n=204: number analyzed (Participants) | 204
  Week 108, n=204 | -2.512 (13.4608)
  Week 120, n=203: number analyzed (Participants) | 203
  Week 120, n=203 | -0.742 (14.3800)
  Week 132, n=205: number analyzed (Participants) | 205
  Week 132, n=205 | -1.499 (13.3816)
  Week 144, n=203: number analyzed (Participants) | 203
  Week 144, n=203 | -0.821 (13.8173)

18. Secondary Outcome: Change From Baseline in Chemistry Parameter: Estimated Glomerular Filtration Rate (eGFR)
Description: Blood samples were collected to analyze the chemistry parameter: eGFR. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Weeks, 12,24,36,48,60,72,84,96,108,120,132,and 144
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
Number analyzed (Participants) | 209
Grams per liter
  Week 12, n=209 | -2.93 (7.250)
  Week 24, n=209 | -1.11 (6.798)
  Week 36, n=209 | -0.63 (7.558)
  Week 48, n=208: number analyzed (Participants) | 208
  Week 48, n=208 | -1.31 (7.378)
  Week 60, n=208: number analyzed (Participants) | 208
  Week 60, n=208 | -0.12 (8.004)
  Week 72, n=208: number analyzed (Participants) | 208
  Week 72, n=208 | 0.84 (7.619)
  Week 84, n=207: number analyzed (Participants) | 207
  Week 84, n=207 | 0.42 (8.731)
  Week 96, n=207: number analyzed (Participants) | 207
  Week 96, n=207 | -0.17 (8.752)
  Week 108, n=205: number analyzed (Participants) | 205
  Week 108, n=205 | 0.42 (8.379)
  Week 120, n=205: number analyzed (Participants) | 205
  Week 120, n=205 | 0.77 (8.826)
  Week 132, n=205: number analyzed (Participants) | 205
  Week 132, n=205 | 0.60 (8.098)
  Week 144, n=204: number analyzed (Participants) | 204
  Week 144, n=204 | 0.95 (8.313)

ADVERSE EVENTS:
Time Frame: On-treatment non-serious adverse events and serious adverse events were collected up to 144 weeks from the start of the treatment
Description: Safety analysis population was used to collect the adverse events
Arm/Group | Tenofovir Disoproxil Fumerate 300 mg
All-Cause Mortality (participants affected / at risk) | 1/213
Serious Adverse Events (participants affected / at risk) | 20/213
Other Adverse Events (participants affected / at risk) | 117/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumerate 300 mg (N=213)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Calculus bladder (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Myocardial bridging (Congenital, familial and genetic disorders) | 1
Adrenal cyst (Endocrine disorders) | 1
Sudden cardiac death (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Epididymal cyst (Reproductive system and breast disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumerate 300 mg (N=213)
Upper respiratory tract infection (Infections and infestations) | 28
Urinary tract infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Anal abscess (Infections and infestations) | 1
Chronic tonsillitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Papilloma viral infection (Infections and infestations) | 1
Pelvic inflammatory disease (Infections and infestations) | 1
Blood creatine phosphokinase increased (Investigations) | 12
Blood uric acid increased (Investigations) | 3
Weight decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Blood phosphorus decreased (Investigations) | 2
Protein urine present (Investigations) | 2
Transaminases increased (Investigations) | 2
Ultrasound liver abnormal (Investigations) | 2
White blood cells urine positive (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Red blood cell count increased (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Chronic gastritis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Reflux gastritis (Gastrointestinal disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 7
Gallbladder polyp (Hepatobiliary disorders) | 3
Hepatic cyst (Hepatobiliary disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic fibrosis (Hepatobiliary disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 3
Steatohepatitis (Hepatobiliary disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 2
Vaginal inflammation (Reproductive system and breast disorders) | 2
Breast hyperplasia (Reproductive system and breast disorders) | 1
Calculus prostatic (Reproductive system and breast disorders) | 1
Prostatic disorder (Reproductive system and breast disorders) | 1
Prostatomegaly (Reproductive system and breast disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 4
Renal cyst (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal injury (Renal and urinary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Achromotrichia acquired (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Insomnia (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Coagulopathy (Blood and lymphatic system disorders) | 2
Splenomegaly (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 4
Arteriosclerosis (Vascular disorders) | 1
Bone formation increased (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Dry eye (Eye disorders) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Visual acuity reduced (Eye disorders) | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Palpitations (Cardiac disorders) | 1
Hamartoma (Congenital, familial and genetic disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bacterial infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT02195518/SAP_000.pdf
  • Study Protocol (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02195518/Prot_001.pdf